CLINICAL TRIAL: NCT00179283
Title: A Multi-center, Randomized, Double-blind, Parallel-group Study of Sertraline vs. Venlafaxine XR in the Acute Treatment of Outpatients With Major Depressive Disorder
Brief Title: Sertraline vs. Venlafaxine XR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Richard C. Shelton, Director of Mood Disorders Clinic, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sert-Ven
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sertraline

INTERVENTIONS:
Drug: sertraline
Drug: venlafaxine XR

SUMMARY:
This is a randomized, double-blind, active control, 8-week, flexible dose study of sertraline vs. venlafaxine Extended Release in the acute treatment of Major Depression in male and female outpatient sites that will recruit 15-20 patients each. Subjects will be randomized in a 1:1 ratio to receive either sertraline or venlafaxine XR based on a computer-generated randomized list.

DETAILED DESCRIPTION:
This is a randomized, double-blind, active control, 8-week, flexible dose study of sertraline vs. venlafaxine XR in the acute treatment of Major Depression in male and female outpatient sites that will recruit 15-20 patients each. Subjects will be randomized in a 1:1 ratio to receive either sertraline or venlafaxine XR based on a computer-generated randomized list.

The primary objectives of the study are: to assess the comparative safety and tolerability of sertraline and venlafaxine XR and to assess number and severity of discontinuation symptoms and time to termination of taper at the end of acute treatment with sertraline vs. venlafaxine XR.

ELIGIBILITY:
Inclusion Criteria:

* Single or Recurrent Episode of MDD without psychotic features
* Additional diagnoses will be permitted only if they are identified as secondary diagnoses
* 18 or above on 17-item Ham-D with item 1 (depressed mood) score of 2 or above

Exclusion Criteria:

* Current or past diagnosis of Bipolar Disorder
* Any history or current psychotic disorder
* Current psychotic symptoms, including current delusional depression
* Current diagnosis of delirium or dementia
* Alcohol or drug abuse or dependence in last 6 months or currently
* Schizoid, Schizotypal, or Borderline Personality Disorder
* Non-response to sertraline at least 150mg for 4 weeks or more, venlafaxine XR at least 225mg for 4 weeks or more, or non-response to 2 antidepressants in the current episode
* Use of any antidepressant within 2 weeks of baseline (4 weeks for fluoxetine)
* Use of herbal and/or homeopathic remedies concomitantly or within 2 weeks of baseline excluding vitamins and mineral supplements
* Use within 1 week of baseline or concomitant use of any psychotropics with the exception zolpidem or zopiclone PRN for sleep
* Use within 4 weeks of baseline of benzodiazepines taken on a regular, daily basis (PRN use is acceptable as long as none in week leading up to randomization)
* Score of 3 or 4 on the suicide item, item 3 of the Ham-D scale at screen or baseline visit
* Participation in any other studies concomitantly or within 90 days prior to entry into this study
* Treatment with monoamine oxidase inhibitors within 14 days of baseline
* Treatment of electroconvulsive therapy within 30 days of baseline
* Previous history or intolerance or hypersensitivity and/or venlafaxine XR
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol
* Presence of serious and/or unstable medical condition
* Abnormal laboratory results
* Positive pregnancy test and/or nursing women or fertile women not practicing an effective method of birth control
* History seizure disorder-excluding febrile seizures of childhood
* Any other condition which in the investigator's judgement might increase the risk to the subject or decrease the chance of obtaining satisfactory data
* Mental condition rendering the subject unable to understand the procedures
* Unable and/or unlikely to comprehend and/or follow the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-04; Study Completion 2003-04

PRIMARY OUTCOMES:
Ham-D (Hamilton Depression Rating Scale for Depression) 17-item
Clinical Global Impression - Severity Scale
Quality of Life, Enjoyment and Satisfaction Questionnaire (Q-LES-Q)
Treatment Emergent Symptom Scale-Revised (TESS-R)
Brief Symptom Inventory (BSI)

SECONDARY OUTCOMES:
NEO-5 factor Inventory (NEO-FFI)
Anxiety Sensitivity Inventory (ASI)
Mood Disorder Questionnaire (MDQ)
Ham-A (Hamilton Rating Scale for Anxiety)
Arizona Sexual Functioning Inventory (A-SEX)
Atypical Features Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Shelton, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Shelton RC, Haman KL, Rapaport MH, Kiev A, Smith WT, Hirschfeld RM, Lydiard RB, Zajecka JM, Dunner DL. A randomized, double-blind, active-control study of sertraline versus venlafaxine XR in major depressive disorder. J Clin Psychiatry. 2006 Nov;67(11):1674-81. doi: 10.4088/jcp.v67n1102. PMID 17196045